CLINICAL TRIAL: NCT00148928
Title: A Multicenter, Open-label Phase I/II Trial to Evaluate the Safety and Activity of CPC-P501 Protein Formulated With the Adjuvant AS15 as First-line Treatment in Patients With Hormone-sensitive Prostate Cancer Who Show Rising PSA
Brief Title: Safety & Activity of P501-AS15 Vaccine as a First-line Treatment for Patients With Hormone-sensitive Prostate Cancer Who Show Rising PSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 102238; 104634
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms, Prostate
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: P501-AS15 vaccine

SUMMARY:
Patients with hormone-sensitive prostate cancer and rising PSA, after primary tumor treatment, will be treated with the P501-AS15 vaccine as out-patients. The maximum dose will be 16 vaccinations, given over a period of approximately one year. Thereafter, the patients' long-term safety and PSA status will be followed over a period of approximately 11 months.

DETAILED DESCRIPTION:
This Phase I/II study will be conducted according to a multicenter, open-label, single-group design at approximately ten centers in Europe. At least 21 HSPC patients with rising PSA after primary tumor treatment will be enrolled in this study. All patients will be treated as out-patients and will receive the same treatment. The maximum dose will be 16 vaccinations. Follow-up: The patients' long-term safety and PSA status will be followed over a period of 48 weeks. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

* Male,
* Aged between 18 and 75 years, inclusive,
* Histologically or cytologically proven adenocarcinoma of the prostate before the initiation of therapy of the primary tumor,
* Radical prostatectomy before progression of disease by rising PSA was established,
* Primary tumor presented a Gleason sum score ≤8,
* Proven progressive hormone-sensitive prostate cancer,
* Serum testosterone level above 50 ng/dl,
* Free of clinically evaluable metastatic disease (other than the rising PSA),
* ECOG Performance Status of 0 or 1,
* Normal organ functions,
* Negative HBV antigen test,
* Negative HCV antibody test,
* The investigator believes that the patient can and will comply with the requirements of the protocol,
* Written, informed consent obtained before enrolment.

Exclusion criteria:

* Orchiectomy,
* Received androgen-deprivation therapy, including neo adjuvant androgen-deprivation therapy,
* Any radiotherapy (external beam radiotherapy and/or brachytherapy) for prostate cancer as primary management,
* Receiving treatment with continuous systemic anticancer medications,
* Received chronic administration of immunosuppressants or other immune-modifying drugs within six months before the first vaccine dose,
* Received any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or the administration of such a product is planned during the study period,
* Receiving any immunoglobulins and/or other blood products or has received such products within the three months preceding the first dose of study vaccine or is planned to receive such products during the study period,
* Received any commercial vaccine within the week before the first study vaccination,
* Previous or concomitant malignancies at other sites, except (i) adequately treated non-melanoma skin cancers, and (ii) effectively treated malignancy that has been in remission for >2 years and is considered by the investigator highly likely to have been cured,
* Any clinical autoimmune disease (except vitiligo),
* Family history of congenital or hereditary immunodeficiency,
* HIV-positive,
* Medical history includes splenectomy or irradiation to the spleen,
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine,
* Any known allergy or hypersensitivity to yeast or yeast products,
* The patient presents with serious acute or chronic illness(es), e.g. active infections requiring antibiotics, bleeding/coagulation disorders, clinically significant heart disease (NCIC CTG III-IV), or other conditions requiring concurrent medications not allowed during this study,
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule,
* History of chronic alcohol consumption and/or drug abuse,
* Acute disease at the time of enrolment. All vaccines can be administered to persons with a minor illness.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2006-11-07 (Actual); Study Completion 2006-11-07 (Actual)

PRIMARY OUTCOMES:
Vaccine-related or possibly vaccine-related Grade 3 or 4 adverse event: a. Any Grade 4 toxicity: fatigue (including lethargy, asthenia, malaise) must have a duration of at least 24 hours. b. Any Grade 3 toxicity with a duration of at least 24 hours | During the study
Clinical PSA response

SECONDARY OUTCOMES:
a. For patients who present a PSA response: The duration of PSA response, The duration of PSA control, The duration of log PSA response. | During the study
b. Humoral immune response induced by P501-AS15 vaccine: Anti-CPC seropositivity. Anti-P501 seropositivity. | At all points during treatment as specified in the study schedule
c. Cellular immune response induced by P501-AS15 vaccine. Frequency of in vitro cellular immune response to CPC P501. | At all points during treatment as specified in the study schedule
d. Any toxicity in terms of solicited symptoms, unsolicited symptoms and serious adverse events. | During the study
e. All adverse events, whether or not associated with toxicity. | During the study
f. General laboratory safety variables. | At all points during treatment as specified in the study schedule

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Turnhout
- France (5):
  - GSK Investigational Site, Auxerre
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villejuif

REFERENCES:
- See also: Results for study 102238 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/102238?search=study&b%22b''%22#rs